CLINICAL TRIAL: NCT02181309
Title: An Open, Randomised, Four-way Crossover Study in Healthy Volunteers to Evaluate the Effect of Food on the Pharmacokinetics of Meloxicam After a Single p.o. Administration of 22.5 mg Meloxicam Oral Suspension and Dose-proportionality Over a Dosage Range of 7.5 mg to 22.5 mg
Brief Title: Effect of Food on the Pharmacokinetics of Meloxicam in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.254
Record Dates: First submitted 2014-07-02; First posted 2014-07-03 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

ARMS (4):
- Meloxicam low dose, fasted (Experimental)
  Interventions: Drug: Meloxicam, low dose
- Meloxicam medium dose, fasted (Experimental)
  Interventions: Drug: Meloxicam, medium dose
- Meloxicam high dose, fed (Experimental)
  Interventions: Drug: Meloxicam, high dose
- Meloxicam high dose, fasted (Active Comparator)
  Interventions: Drug: Meloxicam, high dose

INTERVENTIONS:
Drug: Meloxicam, low dose
  Arms: Meloxicam low dose, fasted
Drug: Meloxicam, medium dose
  Arms: Meloxicam medium dose, fasted
Drug: Meloxicam, high dose
  Arms: Meloxicam high dose, fasted; Meloxicam high dose, fed

SUMMARY:
Study to investigate dose-proportionality over the dosage range 7.5 mg to 22.5 mg, and to assess the effect of food on the pharmacokinetics of meloxicam after a single p.o. administration of 22.5 mg meloxicam oral suspension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Age range from 21 to 50 years
* Broca index +/- 20%
* Written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG and laboratory value) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than ten half-lives of the respective drug prior to administration
* Use of any drugs which might influence the results of the trial (≤ one week prior to administration or during trial)
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range or clinical relevance
* History of haemorrhagic diatheses
* History of gastrointestinal ulcer, perforation or bleeding
* History of bronchial asthma

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. sterilisation, intrauterine pessary, oral contraceptives
* Inability to maintain this adequate contraception during the whole study period
* Lactating

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-01; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Maximum drug plasma concentration (Cmax) | up to 96 hours after drug administration
Total area under the plasma concentration-time curve from time to administration to infinity (AUC0-infinity) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | up to 96 hours after drug administration
Total area under the plasma drug concentration-time curve from time of administration to the last quantifiable drug (AUC0-tf) | up to 96 hours after drug administration
Apparent terminal elimination rate constant (λz) | up to 96 hours after drug administration
Apparent terminal half-life (t1/2) | up to 96 hours after drug administration
Mean total residence time (MRTtot) | up to 96 hours after drug administration
Total clearance, divided by f (CL/f) | up to 96 hours after drug administration
Apparent volume of distribution during the terminal phase, divided by f (Vz/f) | up to 96 hours after drug administration
Number of patients with adverse events | up to 67 days